CLINICAL TRIAL: NCT05730088
Title: The Effect of Post-Discharge Multiple Nursing Interventions on the Number of Hospital Admissions, Dyspnea Level, and Quality of Life in COPD Patients Receiving Home Oxygen Therapy: A Randomized Controlled Study
Brief Title: Reducing the Number of Hospital Admissions With Multiple Nursing Interventions in COPD Patients Using Oxygen Concentrators at Home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Hasan Bakır, lecturer, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NEU-HF-HBAKIR-01
Record Dates: First submitted 2023-01-25; First posted 2023-02-15 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; home visit; multiple nursing intervention; life quality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Interviews as Topic

STUDY DESIGN:
Intervention Model Description: The Effect of Post-Discharge Multiple Nursing Interventions on the Number of Hospital Admissions, Dyspnea Level, and Quality of Life in COPD Patients Receiving Home Oxygen Therapy: A Randomized Controlled Study
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Within the scope of the pre-test, the researcher to the patients who will explain the purpose of the research and agree to participate in the research; Inclusion Criteria Form; Socio-Demographic Information Form; Patient Descriptive Information Form, Modified British Medical Research Council (MRC) Questionnaire, St George Respiratory Questionnaire (Quality of Life Scale) will be used to evaluate patients' symptoms. In addition, the patients in the intervention group will be educated with the training booklet "Educational Guide for COPD Patients" prepared by the researcher by scanning the literature.
  Interventions: Other: health education; Other: Mobile application (Creating a WhatsApp group):; Other: Telephone interview:
- Not intervention group (No Intervention): The control group will be subjected to the standard COPD training given in the hospital and no intervention will be made by the researcher. After the trials of the experimental group are completed, the control group will be given a home visit, a COPD training booklet, and audio-visual materials.

INTERVENTIONS:
Other: health education — Health Education: While they are still in the hospital, a 30-minute individually planned education about their disease will be given to patients using the COPD patient education booklet. step 1. Smoking cessation, step 2. Vaccination, step 3. Correct drug use, step 4. Regular exercise, step 5. Healthy eating, step 6. Coping with stress, step 7 Coping with attacks, step 8. Includes regular oxygen therapy. Let's learn nhaverug treatments in coping with COPD, under the title of pulmonary rehabilitation (Respiratory Rehabilitation), methods of coping with shortness of breath, indoor air pollution and outdoor air pollution subheadings.
  Arms: intervention group
Other: Mobile application (Creating a WhatsApp group): — A group will be created through the WhatsApp application for participants in health education and visual and audio materials will be shared through this group every week. In the coming weeks, the researcher will provide consultancy services to those who have problems with the application.
  Arms: intervention group
Other: Telephone interview: — Participants will be called every month by the researcher and asked if there are any hospital visits in that month, especially if they are chest disease visits.
  Arms: intervention group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a progressive lung disease characterized by persistent airflow obstruction and chronic respiratory symptoms or alpha-1-antitrypsin deficiency in response to inhaled cigarette smoke or other irritants. The excessive morbidity and mortality associated with COPD acute exacerbations represent a significant public health problem that places a high burden on patients, their families and society. In frequent and severe exacerbations, patients may experience a decrease in quality of life, depression, and even death up to one year after hospitalization. Costs associated with COPD are more than $15.5 billion, and hospitalizations and repeated hospital admissions related to acute exacerbations alone account for 70% of all costs. For these reasons, efforts to reduce hospital admissions and hospitalizations associated with recurrent exacerbations are imperative to improve patient's quality of life and reduce the societal burden.

DETAILED DESCRIPTION:
The patients in the intervention group will be called by the researcher within 3-7 days after discharge for the purpose of getting to know each other. The researcher will inform the participants/relatives about the purpose of the study and the procedures to be performed. The date and time for the next call will be given and the next phone call will be planned. The researcher will inform the patients/relatives about the materials sent. During the phone call, any questions the patient has about their illness, medications, or oxygen concentrator will be answered by the researcher. Then, the patient will be asked whether they have been to the hospital after being discharged and this self-reported information will be recorded on the prepared hospital application form. If they have applied to the hospital, the department(s) will be asked and noted. At the end of the phone call, the time and day of the next call will be planned with the patient/relatives. The second phone call will be made by the researcher within 3 months after discharge to the patients in the intervention group and the date and time of the phone call will be planned after the approval of the researcher and the patient/relatives and the call plan will be made. During the phone call, the researcher will first introduce himself/herself and briefly explain why the phone call is being made. During the phone call, any questions the patient may have about his/her illness, medications, or oxygen concentrator will be answered by the researcher. Then, after the patient is discharged, the patient's hospital application will be asked and the answers received based on self-reporting will be written on the hospital application form. If there is a hospital application, the department/departments will be asked and noted. 5 minutes of the phone call will include introductions and general topics about the illness, the second 5 minutes will answer any questions the patient/relatives may have, and the last 5 minutes will end with the researcher providing consultancy services on what needs to be done in the future. Care will be taken not to exceed 20 minutes. At the end of the call, the date and time of the last call will be determined by talking to the patient/relative. In the phone call in the third month, the mMRC dyspnea scale and the St George Respiratory Questionnaire (Quality of Life Scale) and Hospital Application Form interim measurements will be collected by a researcher outside the study.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with stage 4 (group D) COPD according to GOLD criteria
* Being 18 years or older,
* Having a video computer, tablet or phone,
* Having an internet connection at home or on the phone,
* Residing in the city centre of Konya,
* Not having a communication problem, such as an inability to understand/speak Turkish, that would prevent participation in the research,
* Being literate,
* Using an oxygen concentrator at home.

Exclusion Criteria:

* Being illiterate,
* Being diagnosed with first, second and third-stage COPD according to GOLD criteria,
* Having another lung disease in addition to COPD (Lung cancer-Asthma, etc.),
* Having physical and/or mental disabilities,
* Being visually impaired and/or hearing impaired,
* Having a communication problem that prevents participation in the research, such as an inability to understand/speak Turkish,
* Having been diagnosed with Covid-19 or having had it in the past,
* Having a psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
number of hospital admissions | At the end of the 1st month.
  Number of hospital admissions
number of hospital admissions | At the end of the 3st month.
  Number of hospital admissions
number of hospital admissions | At the end of the 6st month.
  Number of hospital admissions

SECONDARY OUTCOMES:
Scores from the mMRC Dyspnea scale (on the first encounter) | At the end of the 1st month.
  0 points for no dyspnea (no respiratory distress when moving quickly on a flat surface or climbing a gentle slope);
  1. point for mild dyspnea (difficulty breathing when moving quickly on a flat surface or climbing a gentle slope);
  2. points for moderate dyspnea (walks slower than peers when walking on level ground, pauses for breathing);
  3. points for severe dyspnea (stopping to breath after walking 100 meters or for a few minutes); and 4 points as very severe dyspnea (shortness of breath while doing daily chores at home, putting on/taking off clothes or going to the toilet).
  As the score increases, the level of dyspnea also increases.
Scores from the mMRC Dyspnea scale (on the first encounter) | At the end of the 3st month.
  0 points for no dyspnea (no respiratory distress when moving quickly on a flat surface or climbing a gentle slope);
  1. point for mild dyspnea (difficulty breathing when moving quickly on a flat surface or climbing a gentle slope);
  2. points for moderate dyspnea (walks slower than peers when walking on level ground, pauses for breathing);
  3. points for severe dyspnea (stopping to breath after walking 100 meters or for a few minutes); and 4 points as very severe dyspnea (shortness of breath while doing daily chores at home, putting on/taking off clothes or going to the toilet).
  As the score increases, the level of dyspnea also increases.
Scores from the mMRC Dyspnea scale (on the first encounter) | At the end of the 6st month.
  0 points for no dyspnea (no respiratory distress when moving quickly on a flat surface or climbing a gentle slope);
  1. point for mild dyspnea (difficulty breathing when moving quickly on a flat surface or climbing a gentle slope);
  2. points for moderate dyspnea (walks slower than peers when walking on level ground, pauses for breathing);
  3. points for severe dyspnea (stopping to breath after walking 100 meters or for a few minutes); and 4 points as very severe dyspnea (shortness of breath while doing daily chores at home, putting on/taking off clothes or going to the toilet).
  As the score increases, the level of dyspnea also increases.
Scores from the St George Respiratory Questionnaire | At the end of the 1st month.
  The total score that can be obtained from the scale is 0 min. - 100 max. The number zero indicates good health, and the number 100 indicates poor health. The scale is Likert type and the questions are in the form of "yes" and "no".
  The symptoms section consists of 8 items and is scored in the range of 0-16 points.
  The activity section consists of 16 items and is scored in the range of 0-32 points.
  The effects of the disease section consists of 26 items and is scored in the range of 0-52 points.
Scores from the St George Respiratory Questionnaire | At the end of the 3st month.
  The total score that can be obtained from the scale is 0 min. - 100 max. The number zero indicates good health, and the number 100 indicates poor health. The scale is Likert type and the questions are in the form of "yes" and "no".
  The symptoms section consists of 8 items and is scored in the range of 0-16 points.
  The activity section consists of 16 items and is scored in the range of 0-32 points.
  The effects of the disease section consists of 26 items and is scored in the range of 0-52 points.
Scores from the St George Respiratory Questionnaire | At the end of the 6st month.
  The total score that can be obtained from the scale is 0 min. - 100 max. The number zero indicates good health, and the number 100 indicates poor health. The scale is Likert type and the questions are in the form of "yes" and "no".
  The symptoms section consists of 8 items and is scored in the range of 0-16 points.
  The activity section consists of 16 items and is scored in the range of 0-32 points.
  The effects of the disease section consists of 26 items and is scored in the range of 0-52 points.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK CİNGİL, Principal Investigator — https://erbakan.edu.tr/hemsirelikfak
Locations (1):
- Selçuk Tıp Fakültesi Hastanesi, Konya, Turkey (Türkiye)